CLINICAL TRIAL: NCT05888623
Title: Computer Assisted Detection of Neoplasia During Colonoscopy Evaluation (CADeNCE)
Brief Title: Computer Assisted Detection of Neoplasia During Colonoscopy Evaluation
Acronym: CADeNCE
Status: Completed | Type: Observational
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason A. Dominitz, MD, MHS, Executive Director, National Gastroenterology and Hepatology Program, VA Puget Sound Health Care System
Other Study IDs: VHA_NGHP_001
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Neoplasms
Keywords: colonoscopy; artificial intelligence; adenoma; Veterans; quality assurance
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Computer Assisted Detection: Colonoscopies performed at a VA facility with computer assisted detection (CADe) artificial intelligence available.
  Interventions: Device: Computer Assisted Detection
- Conventional Colonoscopy: Colonoscopies performed at a VA facility without CADe artificial intelligence available

INTERVENTIONS:
Device: Computer Assisted Detection — Computer-assisted polyp detection system that utilizes artificial intelligence (AI) during colonoscopy
  Other Names: GI Genius Intelligent Endoscopy Module (Medtronic)
  Groups: Computer Assisted Detection

SUMMARY:
The goal of this cluster randomized study is to determine if artificial intelligence systems used during colonoscopy can improve the detection of precancerous polyps in the colon. The primary question it aims to answer is whether computer-assisted detection devices improve the proportion of colonoscopies found to have precancerous adenomatous polyps.

Secondary aims will assess if computer-assisted detection devices improve the proportion of colonoscopies found to other types of precancerous polyps known as sessile serrated lesions, or cancer of the colon and rectum. The study will also assess possible negative effects of use of computer-assisted detection (e.g., prolonging the procedure time or false-positive biopsies) and survey device users to learn about their experience with this technology.

The study team will provide computer-assisted detection devices to randomly chosen VA medical centers for use during colonoscopy and compare colonoscopy findings for patients who undergo colonoscopy at facilities that are equipped with these devices to the findings of patients who undergo colonoscopy at VA facilities that do not have these devices.

A survey will be distributed to physicians who perform colonoscopy to assess their experience using computer-assisted detection devices.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy performed at a Veterans Affairs (VA) medical center

Exclusion Criteria:

* Colonoscopy performed at VA medical centers that acquired computer-assisted detection artificial intelligence devices through non-random assignment
* Colonoscopy performed at a VA medical center where pathology results are not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Veterans undergoing colonoscopy for any indication at VA facilities across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 334200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | Baseline and 6 months
  Change in the proportion of colonoscopies in which one or more adenomas are detected

SECONDARY OUTCOMES:
Adenocarcinoma detection rate | Baseline and 6 months
  Change in the proportion of colonoscopies where colorectal cancer is detected
Sessile serrated lesion detection rate | Baseline and 6 months
  Proportion of colonoscopies with one or more sessile serrated lesions detected
Proportion of colonoscopies with pathology obtained | Baseline and 6 months
  Proportion of colonoscopies where specimens were obtained for pathologic review
Proportion of pathology without adenoma or adenocarcinoma | Baseline and 6 months
  As a surrogate for false positive lesion identification during use of CADe
Withdrawal time without interventions | Baseline and 6 months
  Change in the duration of colonoscope withdrawal when no intervention (e.g., polypectomy, biopsy) is performed. This outcome can only be assessed at a subset of sites due to data availability issues (i.e., Provation MD sites).
Provider satisfaction with computer assisted detection for colonoscopy | Approximately 6 months after deployment
  Provider ratings of satisfaction with the CADe device

CONTACTS AND LOCATIONS:
Overall Officials: Jason A. Dominitz, MD, MHS, Study Director — US Department of Veterans Affairs
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy I, Bruckmayer L, Klang E, Ben-Horin S, Kopylov U. Artificial Intelligence-Aided Colonoscopy Does Not Increase Adenoma Detection Rate in Routine Clinical Practice. Am J Gastroenterol. 2022 Nov 1;117(11):1871-1873. doi: 10.14309/ajg.0000000000001970. Epub 2022 Aug 23. PMID 36001408
- [Background] Ladabaum U, Shepard J, Weng Y, Desai M, Singer SJ, Mannalithara A. Computer-aided Detection of Polyps Does Not Improve Colonoscopist Performance in a Pragmatic Implementation Trial. Gastroenterology. 2023 Mar;164(3):481-483.e6. doi: 10.1053/j.gastro.2022.12.004. Epub 2022 Dec 15. No abstract available. PMID 36528131
- [Background] Wallace MB, Sharma P, Bhandari P, East J, Antonelli G, Lorenzetti R, Vieth M, Speranza I, Spadaccini M, Desai M, Lukens FJ, Babameto G, Batista D, Singh D, Palmer W, Ramirez F, Palmer R, Lunsford T, Ruff K, Bird-Liebermann E, Ciofoaia V, Arndtz S, Cangemi D, Puddick K, Derfus G, Johal AS, Barawi M, Longo L, Moro L, Repici A, Hassan C. Impact of Artificial Intelligence on Miss Rate of Colorectal Neoplasia. Gastroenterology. 2022 Jul;163(1):295-304.e5. doi: 10.1053/j.gastro.2022.03.007. Epub 2022 Mar 15. PMID 35304117
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963
- [Background] Gawron AJ, Yao Y, Gupta S, Cole G, Whooley MA, Dominitz JA, Kaltenbach T. Simplifying Measurement of Adenoma Detection Rates for Colonoscopy. Dig Dis Sci. 2021 Sep;66(9):3149-3155. doi: 10.1007/s10620-020-06627-2. Epub 2020 Oct 8. PMID 33029706

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT05888623/Prot_SAP_000.pdf